CLINICAL TRIAL: NCT05623956
Title: Circulating Metabolites and Tumor-derived Extravesicular Proteins in Small Cell Lung Cancer
Brief Title: Proteomics in Small Cell Lung Cancer
Acronym: SCLC-OMICS
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Weronika Maria Szejniuk, MD, PhD, Aalborg University Hospital
Other Study IDs: N-20220023
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Cancer
Keywords: Proteomics; Biomarkers
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to gather insight into tumor-derived circulating extracellular vesicles-proteins in patients with newly diagnosed small cell lung cancer.

DETAILED DESCRIPTION:
The study will include 50 patients with newly diagnosed SCLC, referred to systemic antineoplastic treatment at the Dept. of Oncology, Aalborg University Hospital and blood samples from 50 healthy blood donors.

The blood samples from SCLC patients will be collected before chemotherapy with Carboplatin and Etoposide and after 2 cycles of chemotherapy.

Imaging will be performed at the Dept. of Radiology, Aalborg University Hospital before chemotherapy and after 3 cycles of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent
* Histopathologically and/or cytologically newly-diagnosed SCLC
* Measurable disease on CT scans
* Eligibility to receive standard chemotherapy consisting of carboplatin and etoposide

Exclusion Criteria:

* Active biopsy-verified second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ
* Prior treatment for any malignant diseases other than non-melanoma skin cancer and cervical carcinoma in situ
* Concomitant anticoagulation treatment (acetylsalicylic acid and clopidogrel are allowed)
* Treatment with any other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 50 patients with newly diagnosed SCLC, referred to systemic antineoplastic treatment at the Dept. of Oncology, Aalborg University Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification and validation of protein biomarkers | 3 years
  For identification and validation of protein biomarkers both untargeted and targeted proteomics will be performed, including a discovery-based bottom-up mass spectrometry approach and label-free Quantification Nano Liquid Chromatography Tandem Mass Spectrometry (LFQ nLC-MS/MS), enzyme-linked immunosorbent assay (ELISA)-based proteomics, and Western Blot analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Weronika Szejniuk, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Region North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No